CLINICAL TRIAL: NCT04999163
Title: Aortix Therapy for Perioperative Reduction of Kidney Injury
Acronym: A Priori
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: It has been decided that further enrollment in this study, as designed, will not be able to answer the proposed hypothesis of the study.
Sponsor: Procyrion (Industry)
Collaborators: Procyrion Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PVP054
Record Dates: First submitted 2021-08-03; First posted 2021-08-10 (Actual); Results first posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-10

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Aortix Arm (Experimental): Subject receives the Aortix device.
  Interventions: Device: Aortix System
- Non-Aortix Arm (No Intervention): Control Arm consists of subjects who choose not to receive the Aortix device or who do not meet the anatomical requirements to receive the Aortix device.

INTERVENTIONS:
Device: Aortix System — Aortix is indicated as a partial circulatory support device to increase renal perfusion and reduce the incidence of acute kidney injury (AKI) in patients undergoing cardiac surgery who are at heightened risk of developing AKI.
  Arms: Aortix Arm

SUMMARY:
The study is a prospective, non-randomized feasibility study to evaluate the safety and performance of providing support with the Aortix System to patients at heightened risk of acute kidney injury (AKI) undergoing cardiovascular surgery.

DETAILED DESCRIPTION:
The study is a prospective, non-randomized feasibility study to evaluate the safety and performance of providing support with the Aortix System to patients at heightened risk of acute kidney injury (AKI) undergoing cardiovascular surgery. Patients who decline Aortix system implant or fail to meet anatomical requirements for Aortix implant will be followed in the non-Aortix arm. Both arms will have the same visit schedule and data collection requirements with the exception of data pertaining to the Aortix system. Data will be reported for both groups.

ELIGIBILITY:
Inclusion Criteria:

1. Have the following risk factor(s) for AKI prior to surgery:

   1. Estimated glomerular filtration rate (eGFR) of ≥ 15 and < 30 ml/min/1.73m2, OR
   2. eGFR ≥ 30 and < 60 ml/min/1.73m2 and ONE or more of the following:

      1. Diabetes (regardless of cause) with metabolic, renal, ophthalmic, neurologic, circulatory, or other complications
      2. Documented NYHA class III or IV heart failure within 1 year prior to enrollment
      3. Left ventricular ejection fraction < 35%
      4. Hypertension with comorbid heart or kidney disease
      5. Persistent Atrial Fibrillation
2. Planned (non-emergency) cardiac surgical procedure including, but not limited to coronary bypass surgery, surgical valve replacement or valve repair
3. Age >21 years, willing and able to provide written informed consent.

   -

Exclusion Criteria:

1. An eGFR of <15 ml/min/1.73m2 at enrollment
2. Cardiac surgical procedure that uses femoral artery cannulation for cardiopulmonary bypass
3. Current support with a durable LVAD, intra-aortic balloon pump, extracorporeal membrane oxygenation (ECMO), or percutaneous ventricular assist devices (e.g., Impella or TandemHeart)
4. Patient has known hypo- or hyper-coagulable state such as disseminated intravascular coagulation or heparin induced thrombocytopenia (HIT)
5. Endovascular procedure with ilio-femoral access >12F within previous 30 days
6. Severe Bleeding Risk (any of the following):

   1. Previous intracranial bleed such that the patient cannot safely use anticoagulation per the study requirements
   2. Platelet count <75,000 cells/mm3
   3. Uncorrectable bleeding diathesis or coagulopathy (e.g., INR ≥ 2 not due to anticoagulation therapy
7. Current endovascular stent graft in the descending aorta or either ilio-femoral vessels
8. Contraindicated Anatomy:

   1. Descending aortic anatomy that would prevent safe placement of the device [<18 mm or >31 mm aorta diameter at deployment location (measured between the superior aspect of the T10 vertebra and superior aspect of the L1 vertebra)]
   2. Ilio-femoral diameter or peripheral vascular anatomy that would preclude safe placement of a 21F (outer diameter) introducer sheath
   3. Abnormalities or severe vascular disease that would preclude safe access and device delivery (e.g., aneurysm with thrombus; marked tortuosity; significant narrowing or inadequate size of the abdominal aorta, iliac, or femoral arteries; or severe calcification)
   4. Known connective tissue disorder (e.g., Marfan Syndrome) or other aortopathy at risk of vascular injury
9. Known hypersensitivity or contraindication to study required medications (e.g., anticoagulation therapy) or device materials (e.g., history of severe reaction to nickel or nitinol)
10. Positive pregnancy test if of childbearing potential
11. Participation in any other clinical investigation that is likely to confound study results or affect the study

    -

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-07-17 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2023-08-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (5):
  - Royal Adelaide Hospital, Adelaide
  - Prince Charles Hospital, Brisbane
  - Princess Alexandra Hospital, Brisbane
  - Monash Health, Melbourne
  - Macquarie University, Sydney

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at 4 investigational sites in Australia between July 17, 2022 and August 7, 2023.
Groups:
- Aortix Arm: Patients who meet all inclusion and none of the exclusion criteria for the study and agree to receive the Aortix system implant are followed in the Aortix Arm.
- Non-Aortix Arm: Patients who decline Aortix system implant or fail to meet anatomical requirements for Aortix implant are followed in the non-Aortix arm.
Period: Overall Study
Arm/Group | Aortix Arm | Non-Aortix Arm
Started | 11 | 9
Completed | 8 | 9
Not Completed | 3 | 0
Not completed — Surgery completed at hospital not participating in the study. | 1 | 0
Not completed — Study enrollment stopped prior to implant. | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants that completed the study follow-up.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aortix Arm | Non-Aortix Arm | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (8.67) | 71.4 (6.98) | 68.9 (8.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 9 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 8 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
AKI Stage [Count of Participants; unit: Participants] — AKI Stage as defined by the Kidney Disease Improving Global Outcomes (KDIGO) clinical practice guidelines to define the level of acute kidney injury. Stage 1 is the lowest level of kidney injury with Stage 3 being the most severe. None refers to no acute injury.
  Participants
    AKI Stage 1 | 1 | 1 | 2
    AKI Stage 2 | 0 | 0 | 0
    AKI Stage 3 | 0 | 2 | 2
    None | 7 | 6 | 13
eGFR [Mean (Standard Deviation); unit: ml/min/1.73m^2] | 49.9 (8.32) | 46.6 (10.82) | 48.1 (9.58)
NYHA Classification [Count of Participants; unit: Participants] — New York Heart Association (NYHA) Classification is used to classify the level of heart failure the subject is currently experiencing. NYHA Class I indicates no physical limitation due to heart failure, Class II indicates mild, Class III indicates moderate and Class IV indicates severe limitations due to heart failure.
  Participants
    Class I | 2 | 3 | 5
    Class II | 0 | 3 | 3
    Class III | 5 | 3 | 8
    Class IV | 1 | 0 | 1
LVEF [Mean (Standard Deviation); unit: percentage of LV ejection fraction] | 47.0 (16.46) | 56.8 (13.24) | 52.2 (15.21)
Height [Mean (Standard Deviation); unit: cm] | 172.6 (8.92) | 172.9 (9.37) | 172.7 (8.87)
Weight [Mean (Standard Deviation); unit: kg] | 101.4 (19.74) | 76.0 (13.31) | 88.0 (20.71)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 32.2 (7.04) | 25.4 (4.05) | 29.1 (6.71)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events Related to Aortix
Description: The number of participants with Serious Adverse Events related to the Aortix implant, retrieval, and therapy.
Time Frame: Enrollment to 30 days post-surgery
Population: All participants that had an attempted or successful Aortix device implant.
Measure: Count of Participants; unit: Participants
Groups:
- Aortix Arm: Participants who meet all the inclusion and none of the exclusion criteria and agree to receive the Aortix device implant.
Arm/Group | Aortix Arm
Number analyzed (Participants) | 8
Participants
  Bleeding (BARC 3b) | 1
  Hemolysis, Transient, Major | 1
  No Serious Related Adverse Events | 6

2. Primary Outcome: Number of Participants With Baseline AKI Stage Compared to AKI Stage at 72 Hours Post-surgery
Description: The intention is to characterize the change in severity of acute kidney injury observed at 72 hours post-surgery using the KDIGO AKI staging criteria. AKI Stage as defined by the Kidney Disease Improving Global Outcomes (KDIGO) clinical practice guidelines defines the level of acute kidney injury with Stage 1 being the lowest level of kidney injury and Stage 3 being the most severe. None refers to no acute kidney injury.
Time Frame: Baseline to 72 hours post-surgery
Population: All participants who completed follow up in the study. 1 participant in the Aortix arm was excluded from analysis due to significant change in medical status.
Measure: Count of Participants; unit: Participants
Arm/Group | Aortix Arm | Non-Aortix Arm
Number analyzed (Participants) | 7 | 9
Participants
  No Change | 1 | 7
  From None to AKI Stage 1 | 4 | 0
  From None to AKI Stage 2 | 1 | 0
  From None to AKI Stage 3 | 1 | 0
  From AKI Stage 1 to None | 0 | 1
  Missing Data | 0 | 1

3. Primary Outcome: Number of Participants Requiring Postoperative Use of Renal Replacement Therapy, Ultrafiltration, and/or Dialysis.
Description: Renal replacement therapy (RRT), ultrafiltration, and dialysis are three treatment options for subjects with severe acute kidney injury and serve as a measure of the degree of acute kidney injury experienced by each group. Any subject receiving any of these therapies prior to 30 days post surgery are counted in this analysis.
Time Frame: Aortix placement to 30 days post- surgery
Population: All participants who completed the study are included in this analysis. One patient in the Aortix Arm was excluded due to significant change in medical status.
Measure: Count of Participants; unit: Participants
Arm/Group | Aortix Arm | Non-Aortix Arm
Number analyzed (Participants) | 7 | 9
Participants | 1 | 1

4. Primary Outcome: Effectiveness
Description: Characterize the rate of 30-day post-surgery readmission due to worsening renal function
Time Frame: If discharged by day 30 post-surgery
Population: Participants who completed the study are included in this analysis. One patient in the Aortix Arm is excluded from this analysis due to significant change in medical status.
Measure: Count of Participants; unit: Participants
Arm/Group | Aortix Arm | Non-Aortix Arm
Number analyzed (Participants) | 7 | 9
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from enrollment to 30-Days post surgery.
Arm/Group | Aortix Arm | Non-Aortix Arm
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 8/8 | 4/9
Other Adverse Events (participants affected / at risk) | 6/8 | 3/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aortix Arm (N=8) | Non-Aortix Arm (N=9)
Hemolysis, Transient, Major (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bleeding (Vascular disorders) | 4 (4) | 2 (2)
Renal Injury (Renal and urinary disorders) | 2 (2) | 1 (1)
Cardiogenic Shock (Cardiac disorders) | 1 (1) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 1 (1)
Vascular Injury (Vascular disorders) | 0 (0) | 1 (1)
Psychiatric Episode (Psychiatric disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Gyn/GU Miscellaneous (Gastrointestinal disorders) | 0 (0) | 1 (1)
Other (General disorders) | 2 (3) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aortix Arm (N=8) | Non-Aortix Arm (N=9)
Renal Injury (Renal and urinary disorders) | 3 (3) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Bleeding Event (Vascular disorders) | 1 (1) | 0 (0)
GI Miscellaneous (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Other (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination of the study leading to small numbers of subjects analyzed. The non-Aortix group did not show the expected incidence of acute kidney injury during and following surgery and therefore a comparison between the groups could not be made. As a result study enrollment was stopped early and the study was terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2022-01-16): https://cdn.clinicaltrials.gov/large-docs/63/NCT04999163/Prot_000.pdf